CLINICAL TRIAL: NCT04771221
Title: Method of Early Diagnosis of Laryngopharyngeal Reflux in an Outpatient Appointment of an Otorhinolaryngologist
Brief Title: Method of Early Diagnosis of Laryngopharyngeal Reflux
Acronym: LPR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kazakh Medical University of Continuing Education (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 14-2020; 14-2020 (Other: KazMUCE)
Record Dates: First submitted 2021-02-23; First posted 2021-02-25 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2022-04

CONDITIONS: Laryngopharyngeal Reflux; Laryngopharyngitis Chronic; Gastro Esophageal Reflux; Laryngitis
Keywords: Laryngopharyngeal Reflux; Laryngopharyngitis Chronic; Gastro Esophageal Reflux; Laryngitis; pH monitoring; pH metric; acoustic voice analysis
MeSH Terms: conditions — Laryngopharyngeal Reflux; Gastroesophageal Reflux; Laryngitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Main group (Experimental): Patients with complaints of sore throat, coughing, burning sensation in the throat, cough, frequent sore throat, difficulty swallowing, lump in the throat, feeling of a foreign body in the throat, voice change, heartburn, belching.
  Interventions: Diagnostic Test: pH metry; Diagnostic Test: Filling out the questionnaire; Device: Endoscopic laryngoscopy; Device: Acoustic voice analysis
- Control group 1 (Experimental): Patients with an early diagnosis of Gastroesophageal reflux disease
  Interventions: Diagnostic Test: pH metry; Diagnostic Test: Filling out the questionnaire; Device: Endoscopic laryngoscopy
- Control group 2 (Experimental): Patients without complaints of sore throat, coughing, burning sensation in the throat, cough, frequent sore throat, difficulty swallowing, lump in the throat, feeling of a foreign body in the throat, voice change, heartburn, belching.
  Interventions: Diagnostic Test: pH metry; Diagnostic Test: Filling out the questionnaire; Device: Endoscopic laryngoscopy

INTERVENTIONS:
Diagnostic Test: pH metry — The collection of mucus from the laryngopharynx to determine the acid-base values through pH-metry.
Diagnostic Test: Filling out the questionnaire — Completion of the questionnaire index of reflux symptoms. An analysis of the results of the effectiveness of this method in patients with complaints of sore throat, coughing, burning sensation in the throat, cough, frequent sore throat, difficulty swallowing, lump in the throat, feeling of a foreign body in the throat, voice change, heartburn, belching will be carried out. Evaluation results range from 0 to 5, where 0 is an indicator of no problem, and 5 is an indicator of a serious problem
Device: Endoscopic laryngoscopy — Video laryngoscopy and assessment of the presence / severity of the symptoms. Evaluation results range from 0 to 4, where 0 is an indicator of no problem, and 4 is an indicator of a serious problem
Device: Acoustic voice analysis — acoustic analysis of the voice was performed in singers with voice disorders before and after treatment using program of the Lingwaves
  Arms: Main group

SUMMARY:
The investigator will issue a Patient Information Consent for the participant in the study. 1.Patients will be asked to complete the Reflux Symptom Index questionnaire.

Clinical survey, medical history. 2. Objective methods for assessing the patient's condition:

- examination of ENT organs. 3. Laboratory and instrumental research methods: Endoscopic laryngoscopy and video laryngoscopy, pH-metry, acoustic voice analysis.

4.Sociological method. 5. Subjective methods for assessing the condition of the larynx. 6. Аnalysis of the received data

DETAILED DESCRIPTION:
The investigator will issue a Patient Information Consent for the participant in the study. 1.Patients will be asked to complete the Reflux Symptom Index questionnaire.

Clinical survey, medical history 2. Objective methods for assessing the patient's condition:

- examination of ENT organs: rhinoscopy, otoscopy, pharyngoscopy and laryngoscopy 3. Laboratory and instrumental research methods - Endoscopic laryngoscopy and video laryngoscopy. pH-metry: The collection of mucus from the laryngopharynx for the determination of acid-base values. Acoustic voice analysis: objective assessment of the voice condition 4.Sociological method: determination of lifestyle, nutrition, the presence or absence of bad habits.

5. Subjective methods for assessing the condition of the larynx - Questionnaires.

6. Аnalysis of the received data

ELIGIBILITY:
Inclusion Criteria:

* Patient's informed consent
* Age: 18-75 years old
* No serious somatic diseases.
* Patients with complaints of sore throat, coughing, burning sensation in the throat, coughing, frequent sore throat, difficulty swallowing, lump in the throat, foreign body feeling in the throat, voice changes, heartburn and belching.
* Diagnosis: Chronic pharyngitis
* Chronic laryngitis

Exclusion Criteria:

* Disagreement to participate in scientific research
* Age: under 18 and over 76
* Severe somatic diseases, organic lesions of the gastrointestinal tract and ENT organs
* Patients with pulmonary pathologies
* Patients with allergic manifestations (seasonal hay fever, asthma, etc.)
* With diagnoses: Acute respiratory diseases
* Patients with general neuralgic disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 385 (Actual)
Dates: Start 2021-01-10 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2022-02-15 (Actual)

PRIMARY OUTCOMES:
Acidity level of the main group, Week 0 | at the inclusion to the study
  The acidity level of the larynx is assessed using litmus paper. The range of acidity levels is from 4.5 to 9.0, where below 6.5 indicates the acidity of the environment, above 7.5 - alkalinity.
Acidity level of the control group 1, Week 0 | at the inclusion to the study
  The acidity level of the larynx is assessed using litmus paper. The range of acidity levels is from 4.5 to 9.0, where below 6.5 indicates the acidity of the environment, above 7.5 - alkalinity.
Acidity level of the control group 2, Week 0 | at the inclusion to the study
  The acidity level of the larynx is assessed using litmus paper. The range of acidity levels is from 4.5 to 9.0, where below 6.5 indicates the acidity of the environment, above 7.5 - alkalinity.
"Index of reflux symptoms" of the main group, Week 0 | at the inclusion to the study
  Patients will be asked to complete the Reflux Symptom Index questionnaire. An analysis of the results of the effectiveness of this method in patients with complaints of sore throat, coughing, burning sensation in the throat, cough, frequent sore throat, difficulty swallowing, lump in the throat, feeling of a foreign body in the throat, voice change, heartburn, belching will be carried out. The severity of the problem is calculated as the summation of all points. The problem is absent if the summation of points is 0. The problem is serious if the summation of points is 5.
"Index of reflux symptoms" of the control group 1, Week 0 | at the inclusion to the study
  Patients will be asked to complete the Reflux Symptom Index questionnaire. An analysis of the results of the effectiveness of this method in patients with complaints of sore throat, coughing, burning sensation in the throat, cough, frequent sore throat, difficulty swallowing, lump in the throat, feeling of a foreign body in the throat, voice change, heartburn, belching will be carried out. The severity of the problem is calculated as the summation of all points. The problem is absent if the summation of points is 0. The problem is serious if the summation of points is 5.
"Index of reflux symptoms" of the control group 2, Week 0 | at the inclusion to the study
  Patients will be asked to complete the Reflux Symptom Index questionnaire. An analysis of the results of the effectiveness of this method in patients with complaints of sore throat, coughing, burning sensation in the throat, cough, frequent sore throat, difficulty swallowing, lump in the throat, feeling of a foreign body in the throat, voice change, heartburn, belching will be carried out. The severity of the problem is calculated as the summation of all points. The problem is absent if the summation of points is 0. The problem is serious if the summation of points is 5.
Endoscopic laryngoscopy of the main group, Week 0 | at the inclusion to the study
  Assessment of the state of the larynx on the scale of reflux symptoms. Where the presence and severity of the sign is assessed in points from 0 to 4. Where 0 is an indicator of no problem, and 4 is an indicator of a serious problem.
Endoscopic laryngoscopy of the control group 1, Week 0 | at the inclusion to the study
  Assessment of the state of the larynx on the scale of reflux symptoms. Where the presence and severity of the sign is assessed in points from 0 to 4. Where 0 is an indicator of no problem, and 4 is an indicator of a serious problem.
Endoscopic laryngoscopy of the control group 2, Week 0 | at the inclusion to the study
  Assessment of the state of the larynx on the scale of reflux symptoms. Where the presence and severity of the sign is assessed in points from 0 to 4. Where 0 is an indicator of no problem, and 4 is an indicator of a serious problem.
Acoustic voice analysis of the main group, Week 0 | at the inclusion to the study
  Acoustic analysis of the voice was performed in patients with a voice profession who had a voice disorder using computer program of the Lingwaves.

SECONDARY OUTCOMES:
Acidity level of the main group, Week 4 | at 4 weeks after initial treatment
  The acidity level of the larynx is assessed using litmus paper. The range of acidity levels is from 4.5 to 9.0, where above 7.5 indicates the alkalinity of the medium, below 6.5 - acidic.
Acidity level of the control group 1, Week 4 | at 4 weeks after initial treatment
  The acidity level of the larynx is assessed using litmus paper. The range of acidity levels is from 4.5 to 9.0, where above 7.5 indicates the alkalinity of the medium, below 6.5 - acidic.
Acidity level of the control group 2, Week 4 | at 4 weeks after initial treatment
  The acidity level of the larynx is assessed using litmus paper. The range of acidity levels is from 4.5 to 9.0, where above 7.5 indicates the alkalinity of the medium, below 6.5 - acidic.
"Index of reflux symptoms" of the main group, Week 4 | at 4 weeks after initial treatment
  Patients will be asked to complete the Reflux Symptom Index questionnaire. An analysis of the results of the effectiveness of this method in patients with complaints of sore throat, coughing, burning sensation in the throat, cough, frequent sore throat, difficulty swallowing, lump in the throat, feeling of a foreign body in the throat, voice change, heartburn, belching will be carried out. The severity of the problem is calculated as the summation of all points. The problem is absent if the summation of points is 0. The problem is serious if the summation of points is 5.
"Index of reflux symptoms" of the control group 1, Week 4 | at 4 weeks after initial treatment
  Patients will be asked to complete the Reflux Symptom Index questionnaire. An analysis of the results of the effectiveness of this method in patients with complaints of sore throat, coughing, burning sensation in the throat, cough, frequent sore throat, difficulty swallowing, lump in the throat, feeling of a foreign body in the throat, voice change, heartburn, belching will be carried out. The severity of the problem is calculated as the summation of all points. The problem is absent if the summation of points is 0. The problem is serious if the summation of points is 5.
"Index of reflux symptoms" of the control group 2, Week 4 | at 4 weeks after initial treatment
  Patients will be asked to complete the Reflux Symptom Index questionnaire. An analysis of the results of the effectiveness of this method in patients with complaints of sore throat, coughing, burning sensation in the throat, cough, frequent sore throat, difficulty swallowing, lump in the throat, feeling of a foreign body in the throat, voice change, heartburn, belching will be carried out. The severity of the problem is calculated as the summation of all points. The problem is absent if the summation of points is 0. The problem is serious if the summation of points is 5.
Endoscopic laryngoscopy of the main group, Week 4 | at 4 weeks after initial treatment
  Assessment of the state of the larynx on the scale of reflux symptoms. Where the presence and severity of the sign is assessed in points from 0 to 4. Where 0 is an indicator of no problem, and 4 is an indicator of a serious problem.
Endoscopic laryngoscopy of the control group 1, Week 4 | at 4 weeks after initial treatment
  Assessment of the state of the larynx on the scale of reflux symptoms. Where the presence and severity of the sign is assessed in points from 0 to 4. Where 0 is an indicator of no problem, and 4 is an indicator of a serious problem.
Endoscopic laryngoscopy of the control group 2, Week 4 | at 4 weeks after initial treatment
  Assessment of the state of the larynx on the scale of reflux symptoms. Where the presence and severity of the sign is assessed in points from 0 to 4. Where 0 is an indicator of no problem, and 4 is an indicator of a serious problem.
Acoustic voice analysis of the main group, Week 4 | at 4 weeks after initial treatment
  Acoustic analysis of the voice was performed in patients with a voice profession who had a voice disorder using computer program of the Lingwaves

CONTACTS AND LOCATIONS:
Overall Officials: Nukusbekova, Principal Investigator — Doctor
Locations (2):
- Kazakhstan (2):
  - SOS Medical Assistance, Almaty
  - V-ent, Almaty

IPD SHARING:
Plan to Share IPD: No